CLINICAL TRIAL: NCT01801917
Title: A Multi-centre Double-blind, Placebo Controlled, Proof of Concept Study to Evaluate the Efficacy and Tolerability of BAF312 in Patients With Polymyositis
Brief Title: Efficacy and Tolerability of BAF312 in Patients With Polymyositis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBAF312X2205
Record Dates: First submitted 2013-02-01; First posted 2013-03-01 (Estimated); Results first posted 2018-01-04 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2018-01

CONDITIONS: Polymyositis
Keywords: Polymyositis; Myositis; PM; chronic muscle inflammation; inflammatory myopathy; inclusion body myositis
MeSH Terms: conditions — Polymyositis; Myositis; Myositis, Inclusion Body | interventions — siponimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): 5 placebo tablets daily during non-titration phase
  Interventions: Drug: Placebo
- BAF312 2mg (Experimental): 1 tablet of BAF312 2 mg + 4 tablets of Placebo daily during non-titration phase
  Interventions: Drug: BAF312
- BAF312 10 mg (Experimental): 5 tablets of BAF312 2 mg daily during non-titration phase
  Interventions: Drug: BAF312

INTERVENTIONS:
Drug: Placebo — Matching placebo tablet for oral administration
  Arms: Placebo
Drug: BAF312 — BAF312 in 4 dosage strengths in tablet form: 0.25 mg, 0.5 mg, 1 mg, 2 mg for oral administration
  Arms: BAF312 10 mg; BAF312 2mg

SUMMARY:
This study assessed the efficacy, safety and tolerability of BAF312 administered orally in patients with clinically active polymyositis and also in patients with polymyositis who had shown inadequate response to corticosteroids and or DMARDs (disease modifying antirheumatic drugs).

DETAILED DESCRIPTION:
This study was stopped prematurely due to overall slow recruitment and no evidence for efficacy in a parallel study in dermatomyositis with an assumed similar pathophysiology. With very small sample sizes per group the overall results for this study including primary and all other efficacy and PD data are inconclusive

ELIGIBILITY:
Inclusion Criteria:

* "definite" or "probable" for polymyositis at least three months before Baseline
* active disease as defined by elevated CK levels, or other enzymes, or MRI/biopsy if enzymes are normal, and persisting muscle weakness
* stable dose of corticosteroid for at least 2 weeks prior to Baseline and should not have received a medium or high dose in the last 8 weeks prior to study entry.
* patients treated with methotrexate must have been on a stable dose for at least 6 weeks prior to Baseline.

Exclusion Criteria:

* Patients with overlap polymyositis, late-stage polymyositis, or other types of myositis.
* Preexisting severe cardiac or pulmonary involvement, malignancy of any organ system or significant eye diseases.
* Uncontrolled diabetes mellitus or diabetes complicated with organ involvement.
* Pregnant or nursing (lactating) women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-04-24 (Actual); Primary Completion 2016-08-05 (Actual); Study Completion 2016-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Novartis Investigative Site, Phoenix, Arizona, United States
- Novartis Investigative Site, Torono, Ontario, Canada
- Novartis Investigative Site, Prague, Czechia
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
- Novartis Investigative Site, Bydgoszcz, Poland
- Novartis Investigative Site, Taichung, Taiwan

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=225

RESULTS

PARTICIPANT FLOW:
Groups:
- BAF312 2mg/BAF312 2mg: Patients in Period 1 continue on same 2 mg dose of BAF312 in Period 2
- BAF312 10 mg/BAF312 10 mg: Patients in Period 1 continue on same 10 mg dose of BAF312 in Period 2
- Placebo/BAF312 2 mg: Patients on placebo in Period 1 switch to active 2 mg BAF312 in Period 2
- Placebo/BAF312 10 mg: Patients on placebo in Period 1 switch to active 10 mg BAF312 in Period 2
Period: Period 1 - Randomized
Arm/Group | BAF312 2mg/BAF312 2mg | BAF312 10 mg/BAF312 10 mg | Placebo/BAF312 2 mg | Placebo/BAF312 10 mg
Started | 7 | 2 | 4 | 1
Completed | 6 | 2 | 3 | 1
Not Completed | 1 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0
Period: Extension - All Active
Arm/Group | BAF312 2mg/BAF312 2mg | BAF312 10 mg/BAF312 10 mg | Placebo/BAF312 2 mg | Placebo/BAF312 10 mg
Started | 6 | 0 | 3 | 0
Completed | 6 | 0 | 3 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BAF312 2mg/BAF312 2mg | BAF312 10 mg/BAF312 10 mg | Placebo/BAF312 2 mg | Placebo/BAF312 10 mg | Total
Number analyzed (Participants) | 7 | 2 | 4 | 1 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (14.78) | 47.0 (21.21) | 48.0 (8.83) | 53.0 (0.0) | 49.4 (12.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 2 | 1 | 10
  Male | 2 | 0 | 2 | 0 | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 7 | 1 | 3 | 0 | 11
  Black | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 1 | 0 | 2
Disease duration [Mean (Standard Deviation); unit: years] | 5.6 (4.46) | 5.4 (2.74) | 2.7 (1.67) | 16.9 (0) | 5.6 (4.77)
Baseline MMT24 Score [Mean (Standard Deviation); unit: scores on a scale] — Manual muscle testing in 24 muscle groups (MMT24). The scores range was 0 to 260. Higher scores indicate better outcome.
  scores on a scale | 202.6 (41.74) | 184.0 (19.80) | 189.5 (45.65) | 166.0 (0) | 193.6 (37.90)
Taking DMARD at baseline [Number; unit: participants] — Taking a disease-modifying antirheumatic drugs
  participants | 7 | 2 | 4 | 1 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 12 for BAF312 2 mg, 10 mg or Placebo (Once Daily) for Combined Efficacy Endpoint: Manual Muscle Testing in 24 Muscles (MMT24)
Description: Manual Muscle Testing Scoring Sheet: Neck flexors, neck extensors and other designated muscles bilaterally (Biceps brachii, Deltoid middle, Quadriceps, Gluteus maximus, Gluteus medius, Trapezius, Iliopsoas, Hamstrings, Wrist extensors, Wrist Flexors, Ankle plantar flexors and Ankle dorsiflexors) were tested on a 0-10 scale by the Investigator. Posterior credibility interval from Bayesian analysis displayed as confidence interval. The scores range was 0 to 260. Higher scores indicate better outcome.
Time Frame: Baseline, at 12 weeks
Population: Pharmacodynamic (PD) included patients with PD data and no major protocol deviations
Measure: Mean (90% Confidence Interval); unit: scores on a scale
Groups:
- BAF312 2mg: 1 tablet of BAF312 2 mg + 4 tablets of Placebo daily during Period 1
- BAF312 10 mg: 5 tablets of BAF312 2 mg daily during Period 1
- Placebo: matching placebo
Arm/Group | BAF312 2mg | BAF312 10 mg | Placebo
Number analyzed (Participants) | 7 | 2 | 5
scores on a scale | 11.2 [3.5 to 19.2] | 39.0 [10.7 to 67.2] | 9.1 [-1.6 to 20.0]
Statistical Analysis 1: Comparison: BAF312 2mg vs Placebo; It was a Bayesian analysis with non-informative prior for co-primary endpoints, MMT-24 and CK, with dual criteria for statistical significance: ≥ 90% posterior probability (PP) of achieving an increase from baseline in MMT24 and decrease in CK and clinical relevance: ≥ 50% PP achieving an increase of 15 points in MMT24 and a decrease of 30% in CK vs. placebo. For this table the value is the posterior probability of achieving an increase in MMT24 and a decrease in CK in 2mg group vs. placebo; Test type: Superiority or Other; Bayesian = 0.586
Statistical Analysis 2: Comparison: BAF312 2mg vs Placebo; It was a Bayesian analysis with non-informative prior for co-primary endpoints, MMT-24 and CK, with dual criteria for statistical significance: ≥ 90% posterior probability (PP) of achieving an increase from baseline in MMT24 and decrease in CK and clinical relevance: ≥ 50% PP achieving an increase of 15 points in MMT24 and a decrease of 30% in CK vs. placebo. . For this table the value is the PP of achieving an increase of 15 points in MMT24 and a decrease of 30% in CK in 2mg group vs. placebo; Test type: Superiority or Other; Bayesian = 0.022
Statistical Analysis 3: Comparison: BAF312 10 mg vs Placebo; It was a Bayesian analysis with non-informative prior for co-primary endpoints, MMT-24 and CK, with dual criteria for statistical significance: ≥ 90% posterior probability (PP) of achieving an increase from baseline in MMT24 and decrease in CK and clinical relevance: ≥ 50% PP achieving an increase of 15 points in MMT24 and a decrease of 30% in CK vs. placebo. For this table the value is the posterior probability of achieving an increase in MMT24 and a decrease in CK in 10mg group vs. placebo; Test type: Superiority or Other; Bayesian = 0.963
Statistical Analysis 4: Comparison: BAF312 10 mg vs Placebo; It was a Bayesian analysis with non-informative prior for co-primary endpoints, MMT-24 and CK, with dual criteria for statistical significance: ≥ 90% posterior probability (PP) of achieving an increase from baseline in MMT24 and decrease in CK and clinical relevance: ≥ 50% PP achieving an increase of 15 points in MMT24 and a decrease of 30% in CK vs. placebo. . For this table the value is the PP of achieving an increase of 15 points in MMT24 and a decrease of 30% in CK in 10mg group vs. placebo; Test type: Superiority or Other; Bayesian = 0.837

2. Primary Outcome: Percent Change From Baseline at Week 12 for BAF312 2 mg, 10 mg or Placebo (Once Daily) Serum Creatine Kinase (CK) Levels
Description: Serum creatine kinase (CK) were analyzed as part of the blood chemistry panel. Posterior credibility interval from Bayesian analysis displayed as confidence interval. The variable CK was log-transformed for statistical analysis and after estimation was converted to percent change from baseline divided by the mean baseline
Time Frame: Baseline, at 12 weeks
Population: Pharmacodynamic (PD) included patients with PD data and no major protocol deviations
Measure: Mean (90% Confidence Interval); unit: U/L
Arm/Group | BAF312 2mg | BAF312 10 mg | Placebo
Number analyzed (Participants) | 7 | 2 | 5
U/L | -19.7 [-32.3 to -4.7] | -55.6 [-77.1 to -13.5] | -0.5 [-21.8 to 25.9]

3. Secondary Outcome: Six-minute Walking Distance (6MWD) at Week 12
Description: This test assessed the distance a patient could walk in 6 minutes (Rutkove et al 2002). If the patient was not able to walk for 6 minutes then a 2 minute walking test was conducted
Time Frame: Baseline, 12 weeks
Population: Pharmacodynamic (PD) included patients with PD data and no major protocol deviations
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | BAF312 2mg | BAF312 10 mg | Placebo
Number analyzed (Participants) | 6 | 1 | 4
meters
  Period 1, Week 12 | 362.47 (52.02) | 393.00 (0.0) | 303.10 (112.480)
  Distance walked,change from BL at Wk 12 | 46.82 (65.64) | 23.00 (0.0) | -6.40 (21.981)

4. Secondary Outcome: Six-minute Walking Distance (6MWD) at Week 24
Description: as for outcome 3
Time Frame: Baseline, 24 weeks
Population: Pharmacodynamic (PD) included patients with PD data and no major protocol deviations
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | BAF312 2mg | Placebo/BAF312 2 mg
Number analyzed (Participants) | 6 | 3
meters
  Period 2, Week 24 | 364.60 (73.803) | 329.33 (186.551)
  Distance walked,change from baseline at Wk 24 | 48.95 (91.922) | 4.33 (51.637)

5. Secondary Outcome: BAF312 Trough Plasma Concentrations (PK Set)
Description: All blood samples were taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein. For each sample, approximately 2 mL of blood was drawn. BAF312 was determined in ethylenediaminetetraacetic acid (EDTA) plasma using a validated liquid chromatography-tandem mass spectrometry (LC-MS/MS) bioanalytical method for the quantification. The anticipated lower limit of quantification (LLOQ) was 0.02 ng/mL using 0.1 mL of plasma
Time Frame: -7 Baseline, day 28, 56, 84
Population: P
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BAF312 2mg | BAF312 10 mg
Number analyzed (Participants) | 6 | 2
ng/mL
  Day - 7 | 0 (0) | 0 (0)
  Day 28: number analyzed (Participants) | 6 | 1
  Day 28 | 25.3 (11.2) | 182 (0)
  Day 56: number analyzed (Participants) | 5 | 1
  Day 56 | 25.1 (12.6) | 270 (0)
  Day 84: number analyzed (Participants) | 6 | 1
  Day 84 | 21.4 (10.1) | 240 (0)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit.
Groups:
- Period 1 BAF312 2mg: Period 1 BAF312 2mg
- Period 1 BAF312 10mg: Period 1 BAF312 10mg
- Period 1 Placebo: Period 1 Placebo
- Period 2 BAF312 2mg/ BAF312 2mg: Period 2 BAF312 2mg/ BAF312 2mg
- Period 2 Placebo/ BAF312 2mg: Period 2 Placebo/ BAF312 2mg
Arm/Group | Period 1 BAF312 2mg | Period 1 BAF312 10mg | Period 1 Placebo | Period 2 BAF312 2mg/ BAF312 2mg | Period 2 Placebo/ BAF312 2mg
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/2 | 0/5 | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 6/7 | 2/2 | 4/5 | 4/6 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1 BAF312 2mg (N=7) | Period 1 BAF312 10mg (N=2) | Period 1 Placebo (N=5) | Period 2 BAF312 2mg/ BAF312 2mg (N=6) | Period 2 Placebo/ BAF312 2mg (N=3)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1 BAF312 2mg (N=7) | Period 1 BAF312 10mg (N=2) | Period 1 Placebo (N=5) | Period 2 BAF312 2mg/ BAF312 2mg (N=6) | Period 2 Placebo/ BAF312 2mg (N=3)
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 0
Feeling cold (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Carbon monoxide diffusing capacity decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Cardiac murmur (Investigations) | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Cerebral artery stenosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 2 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.